CLINICAL TRIAL: NCT00900198
Title: Tissue Procurement Protocol for the Developmental Therapeutics Clinic, National Cancer Institute (NCI)
Brief Title: Collection of Tissue Samples for Cancer Research
Status: Recruiting | Type: Observational
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 060213; 06-C-0213
Record Dates: First submitted 2009-05-09; First posted 2009-05-12 (Estimated); Last update posted 2025-11-28 (Actual); Status verified 2025-07-09

CONDITIONS: Neoplasms; Lymphomas; Multiple Myeloma; Myelodysplastic Syndrome
Keywords: Tissue Collection; Biospecimen; Assay Development; Tissue Acquisition; Tissue Biopsies; Natural History
MeSH Terms: conditions — Neoplasms; Lymphoma; Multiple Myeloma; Myelodysplastic Syndromes | interventions — Biopsy

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Other
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- 1/Standard: Standard
  Interventions: Procedure: Biopsy
- 2/Standard and Preclinical Models: Standard and Preclinical Models
- 3/Preclinical Models: Preclinical Models
- 4/Preclinical Models, Pediatric: Preclinical Models, Pediatric

INTERVENTIONS:
Procedure: Biopsy — Tissue samples will be collected for research purposes from non-surgical procedures, such percutaneous biopsies for the sole purpose of obtaining specimens or biological fluids for the protocol.
  Groups: 1/Standard

SUMMARY:
Background:

-Patients who are being evaluated and/or treated at the NIH Clinical Center and adult patients at participating sites will be entered onto this tissue procurement protocol for collection of tissue specimens.

Objectives:

* To obtain samples from adult and pediatric patients for research purposes from tests and procedures that are done as required by the primary research protocol(s) to which a patient is enrolled or as part of their standard-of-care treatment.
* To obtain samples for research purposes from non-surgical procedures, such as percutaneous biopsies, performed for the sole purpose of obtaining tissue specimens or biological fluids for this protocol.

Eligibility:

-Adult patients (18 years of age and older) and pediatric patients (younger than 18 years of age) who are being evaluated for and/or treated for cancer at the NIH Clinical Center participating sites.

Design:

* This is a multicenter tissue procurement protocol with NCI as the coordinating center.
* For adult patients: specimens for research purposes, as outlined in this protocol, will be obtained from tests and procedures that are done as required by the primary research protocols to which a patient is enrolled or as part of their standard-of-care treatment. Non-surgical procedures, such as percutaneous biopsies, may also be performed for the sole purpose of obtaining tissue specimens or biological fluids for this protocol. Tissues and biological fluids to be procured may include but are not limited to blood, serum, urine, tumor tissue, normal tissue, pleural fluid, CSF, saliva, bronchial alveolar lavage (BAL), circulating tumor cells, hair follicles, and bone marrow. These specimens will be stored with unique identifiers and used to perform only those research studies that are outlined in this protocol.
* For pediatric patients: tumor biopsy/resection tissue used for pediatric preclinical model development will only be from tissue already being obtained as part of a procedure necessary for the patient s clinical care or as part of a primary research protocol; blood specimens will be collected as part of a blood collection already scheduled for the patient s clinical care or as part of the planned pre-procedure bloodwork; volumes collected will not exceed institutional research limits.
* Given the risks associated with any invasive procedure, such as tumor biopsy, the procedure will be discussed in detail with the patients and their parents/guardian (as indicated), including the side effects, prior to obtaining a separate consent for each procedure. A separate consent will not be signed prior to obtaining samples by minimally invasive measures, such as venipuncture.
* This study has two separate consent forms at the NIH Clinical Center: one for adult patients to donate specimens for ongoing research on assay development and studies of molecular pathways, and one for adult and age-appropriate pediatric patients to donate samples for the generation of preclinical models. The study also has consent form templates for adult and pediatric patients at participating sites to donate specimens to create preclinical models.
* Patients may remain on study for the duration of their consent or completion of the planned procedure, whichever comes first.

DETAILED DESCRIPTION:
Background:

Patients who are being evaluated and/or treated at the NIH Clinical Center and at participating sites will be entered onto this tissue procurement protocol for collection of tissue specimens.

Objectives:

To obtain specimens from adult and pediatric patients for research purposes from tests and procedures that are done as required by the primary research protocol(s) to which a patient is enrolled or as part of their standard-of-care treatment.

To obtain specimens for research purposes from non-surgical procedures, such as percutaneous biopsies, performed for the sole purpose of obtaining tissue specimens or biological fluids for this protocol.

Eligibility:

Adult patients (18 years of age and older) and pediatric patients (younger than 18 years of age) who are being evaluated for and/or treated for cancer at the NIH Clinical Center and at participating sites.

Design:

This is a multicenter tissue procurement protocol with NCI as the coordinating center.

For adult patients: specimens for research purposes, as outlined in this protocol, will be obtained from tests and procedures that are done as required by the primary research protocol(s) to which a patient is enrolled or as part of their standard-of-care treatment. Non-surgical procedures, such as percutaneous biopsies, may also be performed on adult patients at the NIH Clinical Center for the sole purpose of obtaining tissue specimens or biological fluids. Tissues and biological fluids to be procured may include blood, serum, urine, tumor tissue, normal tissue, pleural fluid, CSF, saliva, bronchial alveolar lavage (BAL), circulating tumor cells (CTCs), hair follicles, bone marrow and bone marrow aspirate. These specimens will be stored with unique identifiers and used to perform only those research studies that are outlined in this protocol.

For pediatric patients: tumor biopsy/resection tissue used for pediatric preclinical model development will only be from tissue already being obtained as part of a procedure necessary for the patient s clinical care or as part of a primary research protocol; blood specimens will be collected as part of a blood collection already scheduled for the patient s clinical care or as part of the planned pre-procedure bloodwork; volumes collected will not exceed institutional research limits.

Given the risks associated with any invasive procedure, such as tumor biopsy, the procedure will be discussed in detail with the patients and their parents/guardian (as indicated), including the side effects, prior to obtaining a separate consent for each procedure. A separate consent will not be signed prior to obtaining specimens by minimally invasive measures, such as venipuncture.

This study has two separate consent forms at the NIH Clinical Center: one for adult patients to donate specimens for ongoing research on assay development and studies of molecular pathways; and one for adult and age-appropriate pediatric patients to donate samples for the generation of preclinical models. The study also has consent form templates for adult and pediatric patients at participating sites to donate specimens to create preclinical models.

Patients may remain on study for the duration of their consent or completion of the planned procedure, whichever comes first.

ELIGIBILITY:
* INCLUSION CRITERIA - ADULT:
* Patients 18 years of age and older who are being evaluated and/or treated for cancer at the NIH Clinical Center or at participating sites:

  * Who have a newly diagnosed malignancy for which they have not yet received treatment, or
  * Who have a previously treated malignancy that is now recurrent or currently progressing on treatment indicated by:

    * radiographic evidence of tumor growth and/or new metastases, or
    * CBC w/differential and/or flow cytometry, or
    * documented evidence by the treating physician of signs/symptoms of clinical disease progression, or
  * Who are currently undergoing treatment and for whom disease response has not yet been assessed,

    ---In this circumstance, specimen collection should occur as distant in time from the most recent drug administration as possible such as after completion of a treatment cycle and immediately prior to initiation of the next cycle.
  * Patients with ongoing partial response (PR) or stable disease (SD) are eligible.

    * For solid tumor diagnoses, confirmation of viable malignancy and/or <90% tumor necrosis, fibrosis, or hemorrhage per the final pathology must be reported to the coordinating site for patients enrolled with ongoing PR or SD at the time of specimen collection.
    * For hematologic malignancies, confirmation of viable malignancy must be reported to the coordinating site per the final flow cytometry report.
* Ability to understand and willingness to sign a written informed consent document indicating their willingness to have their tissue or biologic fluid specimens used for research as outlined in this protocol.

At the NIH Clinical Center ONLY:

* At the PIs discretion, specimens may be collected from patients 18 years of age and older prior to the development of an invasive cancer, who are being evaluated and/or treated for a confirmed familial cancer syndrome such as but not limited to Hereditary Breast and Ovarian Cancer (HBOC), Hereditary Non-polyposis Colorectal Cancer Syndrome or Hereditary Diffuse Gastric Cancer (HDGC) syndrome.
* Specimens, including blood only, can be collected from patients 18 years of age and older who are being evaluated and/or treated for a hematologic malignancy, including Myelodysplastic Syndrome (MDS) and/or MDS Myeloproliferative Neoplasm (MDS-MPN), that meet all other adult eligibility criteria.

  * Due to the different characteristics of hematologic malignancies versus solid tumor malignancies, including methodology for assessment of disease response, residual disease, and progression, evaluation of these factors for determination of protocol eligibility should be made utilizing established standards such as hematopathology, flow cytometry, immunohistochemical analysis, etc.

EXCLUSION CRITERIA:

Note: Testing for bloodborne pathogens or other infections is not required for eligibility assessment and will be performed only if clinically indicated. Exclusion criteria for bloodborne pathogens and/or other infections is based on existing documentation in the medical record or patient report of such diagnosis at the time of eligibility assessment, if testing is not obtained for clinical indications.

* Patients with cancer-like syndromes and/or blood disorders such as but not limited to systemic mastocytosis, Langerhans cell histiocytosis, chronic eosinophilic leukemia/hypereosinophilic syndrome, lymphomatoid granulomatosis, or monoclonal gammopathy of undetermined significance (MGUS).
* Patients with invasive fungal infections.
* Patients with active and/or uncontrolled infections or who are still recovering from an infection:

  * All antibiotics, antifungals, or antivirals prescribed for the treatment of an infection should be completed at least 1 week (7 days) prior to collection.
  * No recurrence of fever or other symptoms related to infection for at least 1 week (7 days) following completion of antibiotics.
  * Patients receiving antibiotics, antifungals, or antivirals for prophylaxis are permissible.
  * Antibiotics being administered topically at a location distant from the planned tissue collection site or eye drops for a localized infection are permissible.
  * Note: Use of antibiotics for prophylaxis is not an exclusion.
* Patients with Human Immunodeficiency Virus (HIV), active or chronic hepatitis (i.e., quantifiable HBV-DNA and/or positive HbsAg, quantifiable HCV-RNA) or known history of HCV or HBV.
* Patients with Hepatitis A as indicated by anti-HAV IgM reactivity

  --Note: Patients that are anti-HAV IgG reactive only are not excluded
* Blood only collections from patients with solid tumors or hematologic malignancy demonstrating partial or stable disease response:

  * Blood will not be collected from patients whose disease demonstrates ongoing partial response or ongoing stable disease given the poor rate of model generation from such specimens.
  * Blood will not be collected from patients between doses within a single treatment cycle.
* Specimen collections from patients with benign tumors including but not limited to desmoid tumors, carcinoma in situ, or ongoing evidence of complete disease response (CR).

INCLUSION CRITERIA - PEDIATRIC:

* Patients younger than 18 years of age and older than 2 months with a histologically or cytologically confirmed diagnosis of cancer (solid tumor or hematologic malignancy) who are being treated for cancer at the NIH Clinical Center or participating clinical sites and who will already be undergoing a clinically necessary medical procedure during which tumor tissue will be resected or needle biopsy tissue or bone marrow aspirate collected. Tissue from neonates will not be collected.
* Ability and willingness to assent to participation, utilizing an explanation that is understandable/age appropriate, as well as receiving parental permission.

At the NIH Clinical Center ONLY

-At the PI s discretion, clinically indicated tissue collections may occur from patients with pediatric tumors that are generally benign but are known to undergo malignant transformation, e.g., neurofibromatosis, osteochondromas, pheochromocytoma, etc.

EXCLUSION CRITERIA - PEDIATRIC:

Note: Testing for bloodborne pathogens or other infections is not required for eligibility assessment and will be performed only if clinically indicated. Exclusion criteria for bloodborne pathogens and/or other infections is based on existing documentation in the medical record or patient report of diagnosis at the time of eligibility assessment, if testing is not obtained for clinical indications.

* Patients with invasive fungal infections
* Patients with active and/or uncontrolled infections or who are still recovering from an infection:

  * Actively febrile patients with uncertain etiology of febrile episode
  * All antibiotics should be completed at least 1 week (7 days) prior to collection
  * No recurrence of fever or other symptoms related to infection for at least 1 week (7 days) following completion of antibiotics
  * Note: Use of antibiotics for prophylaxis is not an exclusion.
* Patients with Human Immunodeficiency Virus (HIV), active or chronic hepatitis (i.e., quantifiable HBV-DNA and/or positive HbsAg, quantifiable HCV-RNA) or known history of HCV or HBV.
* Patients with Hepatitis A as indicated by anti-HAV IgM reactivity

  --Note: Patients that are anti-HAV IgG reactive only are not excluded
* Specimen collections from patients with benign tumors including but not limited to desmoid tumors, carcinoma in situ, or ongoing evidence of complete disease response (CR) based on imaging.
* Blood only collections from patients with partial or stable disease response:

  * Blood will not be collected from patients whose disease demonstrates ongoing partial response or ongoing stable disease given the poor rate of model generation from such specimens.
  * Blood will not be collected from patients between doses within a single treatment cycle.

Min Age: 2 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients who are being evaluated and/or treated at the NIH Clinical Center (pediatric and adult) and adult patients at participating sites will be entered onto this tissue procurement protocol for collection of tissue specimens
Sampling Method: Non-Probability Sample
Enrollment: 5000 (Estimated)
Dates: Start 2006-07-06 (Actual)

PRIMARY OUTCOMES:
Collection of research samples | Day of collection
  Delinking of patient samples for research

CONTACTS AND LOCATIONS:
Overall Officials: James H Doroshow, M.D., Principal Investigator — National Cancer Institute (NCI)
Locations (17):
- United States (16):
  - UC Davis, Sacramento, California
  - University of Colorado, Denver, Aurora, Colorado
  - Emory University, Atlanta, Georgia
  - Indiana University - Purdue, Indianapolis, Indiana
  - University of Iowa, Iowa City, Iowa
  - Johns Hopkins University, Baltimore, Maryland
  - National Institutes of Health Clinical Center, Bethesda, Maryland
  - University of Michigan Ann Arbor, Ann Arbor, Michigan
  - Washington University - St. Louis, St Louis, Missouri
  - Roswell Park Cancer Institute, Buffalo, New York
  - Ohio State University, Columbus, Ohio
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania
  - Medical University of South Carolina, Charleston, South Carolina
  - University of Utah, Salt Lake City, Utah
  - University of Virginia, Charlottesville, Charlottesville, Virginia
  - Fred Hutchinson, Seattle, Washington
- Princess Margaret Hospital Cancer Centre, Toronto, Canada

REFERENCES:
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?A_2006-C-0213.html